CLINICAL TRIAL: NCT05408819
Title: A Prospective Study on Accuracy and Safety of Coplanar Template Assisted CT-guided Abdominal Tumor Biopsy and Fiducial Marker Implantation
Brief Title: Accuracy of Coplanar Template Assistance for Abdominal Tumor Puncture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Qiu Bin, Principal Investigator, Peking University Third Hospital
Other Study IDs: ChiECRCT20220035
Record Dates: First submitted 2022-05-22; First posted 2022-06-07 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Abdominal Tumor
Keywords: abdominal tumor; biopsy; fiducial marker; coplanar template
MeSH Terms: conditions — Abdominal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coplanar Template group: Paticipant will undergo coplanar template assisted CT-guided abdominal tumor biopsy or fiducial markers implantation and the prospective accuracy and safety data will record.

SUMMARY:
In recent years, template guidance has been applied and developed in the field of puncture related operations, such as template-assisted radioactive seed implantation. With the guidance of template, needle pathway of seed implantation, biopsy and fiducial marker implantation can be precisely planned actual operation, which is conducive to the accurate proceeding. Templates can be divided into coplanar templates and non-coplanar templates. The digital coplanar template coordinate puncture system has been developed in China and has been applied in clinical practice.

In our previous studies, coplanar template assisted CT-guided radioactive seed implantation has good clinical feasibility for percutaneous biopsy of small pulmonary nodules. However, the accuracy of coplanar template assistance for abdominal tumor puncture are lacking in prospective studies. The study aims to prospectively observe the accuracy and safety of coplanar template assisted CT-guided abdominal tumor puncture during biopsy and fiducial markers implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 85
2. Single or multiple abdominal tumors or mass (solid, partially solid)
3. Without taking drugs affecting coagulation and/or platelet aggregation are used; If used, the drug has been discontinued for a sufficient period of time (e.g. 1 week)
4. KPS>60 points, no serious or uncontrolled underlying diseases, clinical evaluation patients can tolerate puncture
5. Planned biopsy and/or fiducial marker implantation with applicable puncture path
6. With informed consent.

Exclusion Criteria:

1. Poor organ function (e.g. lung function FEV1<40% and/or DLCO<50%)
2. The lesion close to blood vessels and intestine, or there is portal vein hypertension and superior vena cava compression, etc., which are expected to have high risks of puncture bleeding and intestinal injury
3. Poor compliance, unable to complete coordination
4. Paticipant who is considered inappropriate or unwilling to participate in this clinical trial for other reasons.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive eligible patient with single or multiple abdominal tumors or mass, who are planned undergo biopsy and/or fiducial marker implantation with applicable puncture path in Peking university Third hospital will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2024-02-10 (Estimated); Study Completion 2024-02-10 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Depth | during the operation
  Depth (millimeter) difference between actual puncture and planned puncture pathway
Accuracy of Angle | during the operation
  Angle (degree) difference between actual puncture and planned puncture pathway

SECONDARY OUTCOMES:
Success rate of needle puncture | during the operation
  Success rate of needle puncture
Complication rate | perioperative the operation
  such as pneumoperitoneum, subcutaneous emphysema, hemorrhage, infection, etc.
operating duration | during the operation
  operating duration from the starting to the ending
Number of CT scans | during the operation
  Number of CT scans

CONTACTS AND LOCATIONS:
Overall Officials: Wang Junjie, Principal Investigator — Peking University Third Hospital
Locations (1):
- Department of Radiation Oncology of Peking university third hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided